CLINICAL TRIAL: NCT01549418
Title: The Risk of Bleeding After Removal of Large Colorectal Polyps in Patients Continuing or Discontinuing on Aspirin: a Multicenter, Double-blind, Placebo-controlled, Randomized Clinical Trial
Brief Title: The Risk of Bleeding After Removal of Large Colorectal Polyps in Patients Taking Aspirin
Acronym: ASAPOL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Jaroslaw Regula, Professor in Gastroenterology, MD, PhD, Maria Sklodowska-Curie National Research Institute of Oncology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ASAPOL
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: Gastrointestinal bleeding; Lower gastrointestinal bleeding (LGIB); Polypectomy; Large colorectal polyps; ASA; Aspirin; Acetylsalicylic acid; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Active Comparator): Patients with at least one large polyps taking aspirin in dose 75 mg daily for 21 days (7 days before and 14 days after polypectomy)
  Interventions: Drug: Aspirin (ASA)
- Placebo (Placebo Comparator): Patients with at least one large polyps taking placebo daily for 21 days (7 days before and 14 days after polypectomy)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin (ASA) — Usage or withdrawal of aspirin (75mg daily per os) 7 days before and 14 days after polypectomy
  Other Names: Not yet named
  Arms: Aspirin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The risk of bleeding after polypectomy of large colorectal polyps in patients taking aspirin is uncertain. This is a randomized, multi-center, placebo-controlled, double-blind study to compare the risk of significant bleeding after endoscopic polypectomy of large (>=10mm) colorectal polyps in patients continuing or discontinuing on daily acetylsalicylic acid (ASA) use. Eligible patients will be randomly assigned in a 1:1 ratio to a group taking 75mg daily ASA or placebo 7 days before and 14 days following polypectomy. The primary endpoint of the study is bleeding within 30 days from colorectal polypectomy. The secondary endpoints are composite cardiovascular events occurring between the date of randomization and 30 days after polypectomy.

DETAILED DESCRIPTION:
Patients chronically taking aspirin (in prophylaxis doses 75-325 mg), with a diagnosis of colorectal polyps ≥ 10 mm in diameter will be enrolled on a routine polypectomy under hospitalization. Meeting the inclusion criteria, after informed consent and a cardiologist consent the patient will receive aspirin/placebo, and The Patient Diary to fill (Visit 1). The patient will be admitted to the Study Center in 6-7 days taking on the aspirin/placebo and prepared for the study (Visit 2). Patient will be under the care of a physician after polypectomy by a minimum of 6 hours. 14 days after polypectomy will be the first control visit, during which the physician will take back patient diary and pack treatment (Visit 3). 30 days after polypectomy will be the second control visit by phone (Visit 4). Patients will be monitored by looking at the end points.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 years or older
2. Daily aspirin for primary or secondary prophylaxis
3. Candidate for endoscopic polypectomy of at least one colorectal polyp 10mm or larger
4. Signed written informed consent
5. Written opinion from a cardiologist that the patient can cease taking aspirin for a period of 21 days in the peri-polypectomy period

Exclusion Criteria:

1. Lifelong anticoagulant therapy with warfarin, acenocumarol
2. Concurrent antiplatelet treatment with clopidogrel or ticlopidin
3. Coagulation disorders INR > 1,5, APTT 2xnorm
4. Known hemorrhagic disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Clinically significant bleeding after colorectal polypectomy | within 30 days after polypectomy
  Clinically significant bleeding after polypectomy - any extravasation of blood from the polypectomy site [immediate (30s after polypectomy), early (to 24ha after polypectomy) or delayed (24ha to 30 days after polypectomy)], with clinical and/or endoscopic and/or laboratory (Hb decline by more than 3 g%)symptoms and would require endoscopic intervention and/or surgical and/or blood transfusions;

SECONDARY OUTCOMES:
Proportion of composite cardiovascular events, ending unplanned hospitalization in both groups aspirin and placebo | in time from randomisation to 30 days after polipectomy
  Composite cardiovascular events - acute coronary syndrome, transient ischemic attack (TIA)or stroke
Proportion of clinically significant delayed bleeding in both groups | within 30 days after polipectomy

CONTACTS AND LOCATIONS:
Overall Officials: Regula Jaroslaw, MD PhD, Study Director — The Medical Centre for Postgraduate Education, and Center of Oncology Institute, Warsaw, Poland; Kaminski F Michal, MD, Study Chair — The Medical Centre for Postgraduate Education, and Center of Oncology Institute, Warsaw, Poland; Pisera Malgorzata, MSc, Principal Investigator — The Medical Centre for Postgraduate Education, and Center of Oncology Institute, Warsaw, Poland